CLINICAL TRIAL: NCT06324864
Title: Testing the Effectiveness of the Culturally Adapted Skills Training START NOW to Reduce Mental Health Problems in Adolescent Refugees
Brief Title: START NOW Adapted: Culturally Adapted Version of START NOW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Christina Stadler (Network)
Responsible Party: Sponsor-Investigator, Prof. Christina Stadler, Prof. Dr. Dr., University Psychiatric Clinics Basel
Organization: University Psychiatric Clinics Basel (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-00212
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Depression; Depression/Anxiety; Anxiety; Adolescent; Emotion Recognition; Mental Health; Resilience,Psychological; Refugee Health
Keywords: randomized controlled trial; effectiveness trial; refugee health; cultural adaptation; skills-training; adolescent migrants
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- START NOW Adapted (Active Comparator): The intervention group will receive a culturally adapted version of the yet well-validated START NOW training. The skills taught within START NOW aim to change dysfunctional negative attitudes and behaviour, improve emotion regulation capacities and enhance the ability to achieve individual goals by addressing key aspects of mental health and resilience. The training includes 10 group sessions including exercises and discussion.
  The sessions will be held by a trained facilitator (staff member of institution, social worker, or else) with the same cultural background in the respective language (depending on group constellation) and supervised by a certified START NOW trainer from the START NOW team.
  Interventions: Behavioral: START NOW Adapted
- Treatment as Usual (No Intervention): The control group will receive treatment as usual.

INTERVENTIONS:
Behavioral: START NOW Adapted — The START NOW skills-training combines aspects of cognitive behavioral therapy (CBT), motivational interviewing (MI), dialectical behavior therapy (DBT), Acceptance and Commitment Therapy (ACT) and trauma-sensitive care. Studies in different contexts have shown START NOW's effectiveness in terms of reducing behavioral problems, reducing hospitalization rates, improving mental health functioning and increasing satisfaction rates. The culturally adapted version will be contextually adapted to different cultural backgrounds and the experience of migration. In ten sessions, participants learn about emotions and are introduced to the START NOW skills. These skills, called "SLOW DOWN", "TAKE A STEP BACK", "ACCEPT", "RESPECT" and "TAKE ACTION", are strategies or techniques that can be used to better manage stress and difficult emotions.
  Arms: START NOW Adapted

SUMMARY:
The goal of this clinical trial is to test the effectiveness of the culturally adapted skills-training START NOW in youth migrant populations. The main question it aims to answer is: Is the culturally adapted skills training START NOW more effective than treatment as usual (TAU) in reducing mental health problems in migrants? Participants will be randomly assigned to the intervention group receiving the skills training START NOW Adapted or the control group receiving TAU. Researchers will compare both groups to see if START NOW Adapted is more effective than TAU in reducing mental health problems in migrants.

DETAILED DESCRIPTION:
Over the last few decades, Europe has experienced one of the largest increases in international migration resulting from a combination of natural and man-made disasters. As these disasters cannot be expected to decrease in the future, it is essential to establish optimal healthcare for migrants, especially refugees. Due to several risk factors of their psychological well-being, refugees have higher prevalence rates of depression, post-traumatic stress disorder (PTSD) and other anxiety disorders compared to the host-country population. Adolescent refugees are particularly vulnerable to mental health problems, as they experience many risk factors associated with their resettlement during crucial phases of their physical and emotional development.

However, despite having a greater healthcare requirement than others, adolescent refugees encounter significant barriers in accessing healthcare services. The skills-training START NOW offers a low-threshold opportunity to treat this vulnerable population by promoting general psychological health and resilience.

Since effective psychological interventions are rooted in a cultural context and must be consistent with clients' cultural beliefs, there is a need to culturally adapt this existing intervention, which has previously been used with Western populations. Our study therefore aims to develop and evaluate a culturally adapted version of the existing START NOW skills-training.

The study is a monocentric, national, confirmatory randomized controlled trial with two arms, namely one intervention and one control group: 1) START NOW Adapted, 2) treatment as usual (TAU). Possible participants taking part in the intervention study are screened for eligibility. For those who are eligible, there will be three assessments: a baseline assessment (t1), a post-treatment assessment (t2), and a 12-weeks follow-up assessment (t3). Randomization into one of the two arms will take place after the baseline assessment (t1) has been conducted. Between t1 and t2, the intervention phase takes place over a period of ten weeks.

ELIGIBILITY:
Inclusion Criteria:

* Being a migrant resettled in Switzerland temporarily or permanently
* Aged between 14 and 18
* Able to speak, read and understand one of the following languages: German, English, Turkish, Farsi, Dari, Ukrainian, Algerian Arabic or Pashto
* Able to give informed consent as documented by signature
* At least sub-clinical depressive symptoms assessed by the Hopkins Symptom Checklist-25 (HSCL-25); total score > 1.75, OR
* Having elevated levels of psychological distress assessed by Kessler Psychological Distress Scale (K10); total score > 20

Exclusion Criteria:

* Suicidality assessed in self-report by the Suicide Behaviors Questionnaire-Revised (SBQ-R; total score > 6) and external report by telephone clarification
* Planning to leave Switzerland in the next 6 months
* Concurrent CBT-based skills-training similar to START NOW

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in symptoms of depression and anxiety at the end of the intervention | From enrollment to the end of treatment at week 14
  Depression and anxiety will be measured by the Hopkins-Symptom-Checklist-25 (HSCL-25) questionnaire. The HSCL-25 is a 25-item self-report questionnaire, on which participants rate if physical, emotional, or psychological symptoms indicating depression, anxiety, and trauma have affected them over the past week. Answers are given on a 4-point Likert Scale (1 = not at all; 4 = extremely), and total scores can range from 25 to 100, with higher scores indicating greater levels of depression, anxiety and trauma, respectively. We chose symptoms of depression and anxiety as the primary endpoint because of their high self-reported prevalence of up to 42% in refugee populations.
Change from baseline in symptoms of depression and anxiety at follow-up | From enrollment to follow-up at week 26
  Depression and anxiety will be measured by the Hopkins-Symptom-Checklist-25 (HSCL-25) questionnaire. The HSCL-25 is a 25-item self-report questionnaire, on which participants rate if physical, emotional, or psychological symptoms indicating depression, anxiety, and trauma have affected them over the past week. Answers are given on a 4-point Likert Scale (1 = not at all; 4 = extremely), and total scores can range from 25 to 100, with higher scores indicating greater levels of depression, anxiety and trauma, respectively. We chose symptoms of depression and anxiety as the primary endpoint because of their high self-reported prevalence of up to 42% in refugee populations.

SECONDARY OUTCOMES:
Change from baseline in self-reported perceived stress at follow-up | From enrollment to follow-up at week 26
  Perceived stress will be measured by the Perceived Stress Scale-10 (PSS-10). The PSS-10 is a 10-item self-report questionnaire including two subscales, on which participants report life as unpredictable, uncontrollable, and overloading over the previous month. Answers are given on a 5-point Likert Scale (0 = never, 4 = very often). Higher scores indicate higher levels of perceived stress. We chose perceived stress as a secondary endpoint because the many pre-, peri- and post-migration stressors that are risk factors for refugees' mental health could be better managed through the intervention aimed at improving distress tolerance.
Change from baseline in self-reported social-ecological resilience at the end of the intervention | From enrollment to the end of treatment at week 14
  Social-ecological resilience will be measured by the Child and Youth Resilience Measure (CYRM-R). The CYRM-R is a 17-item self-report questionnaire measuring resilience that has been validated in 11 different countries. Items include social integration and support, autonomy and fair treatment and can be answered on a 3- point Likert Scale (1 = no, 3 = yes). Higher scores hereby indicate more available protective factors and higher social-ecological resilience. We chose this secondary endpoint because it has often been used to assess the effectiveness of interventions in pre-post and longitudinal designs.
Change from baseline in self-reported perceived stress at the end of the intervention | From enrollment to the end of treatment at week 14
  Perceived stress will be measured by the Perceived Stress Scale (PSS-10). The PSS-10 is a 10-item self-report questionnaire including two subscales, on which participants report life as unpredictable, uncontrollable, and overloading over the previous month. Answers are given on a 5-point Likert Scale (0 = never, 4 = very often). Higher scores indicate higher levels of perceived stress. We chose perceived stress as a secondary endpoint because the many pre-, peri- and post-migration stressors that are risk factors for refugees' mental health could be better managed through the intervention aimed at improving distress tolerance.
Change from baseline in self-reported social-ecological resilience at follow-up | From enrollment to the end of treatment at week 14
  Social-ecological resilience will be measured by the Child and Youth Resilience Measure (CYRM-R). The CYRM-R is a 17-item self-report questionnaire measuring resilience that has been validated in 11 different countries. Items include social integration and support, autonomy and fair treatment and can be answered on a 3- point Likert Scale (1 = no, 3 = yes). Higher scores hereby indicate more available protective factors and higher social-ecological resilience. We chose this secondary endpoint because it has often been used to assess the effectiveness of interventions in pre-post and longitudinal designs.
Change from baseline in facial emotion recognition at the end of the intervention | From enrollment to the end of treatment at week 14
  Facial emotion recognition will be measured using the Penn Emotion Recognition Task (ER-40). The ER-40 consists of 40 colour photographs of static multicultural faces expressing four basic emotions (i.e. happiness, sadness, anger or fear) and neutral expressions. Participants quickly select the appropriate emotion label for each face. They then rate their confidence in the accuracy of their response on a scale from 0 (not at all confident) to 100 (extremely confident). Accuracy scores range from 0 to 40. The ER-40 has strong psychometric properties and is recommended for use in clinical trials. We included the secondary endpoint facial emotion recognition (ER) as performance on measures of emotion recognition is a first step in emotion regulation.
Change from baseline in facial emotion recognition at follow-up | From enrollment to follow-up at week 26
  Facial emotion recognition will be measured using the Penn Emotion Recognition Task (ER-40). The ER-40 consists of 40 colour photographs of static multicultural faces expressing four basic emotions (i.e. happiness, sadness, anger or fear) and neutral expressions. Participants quickly select the appropriate emotion label for each face. They then rate their confidence in the accuracy of their response on a scale from 0 (not at all confident) to 100 (extremely confident). Accuracy scores range from 0 to 40. The ER-40 has strong psychometric properties and is recommended for use in clinical trials. We included the secondary endpoint facial emotion recognition (ER) as performance on measures of emotion recognition is a first step in emotion regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Janine Bacher, MSc, Principal Investigator — University Psychiatric Clinics Basel
Locations (1):
- University Psychiatric Clinics Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bacher J, Stadler C, Unternaehrer E, Brunner D. Testing the effectiveness of the culturally adapted skills training START NOW to reduce mental health problems in adolescent refugees: study protocol for a randomized controlled trial. Front Public Health. 2024 Jun 11;12:1408026. doi: 10.3389/fpubh.2024.1408026. eCollection 2024. PMID 38919921
- [Background] Stadler C, Freitag CM, Popma A, Nauta-Jansen L, Konrad K, Unternaehrer E, Ackermann K, Bernhard A, Martinelli A, Oldenhof H, Gundlach M, Kohls G, Pratzlich M, Kieser M, Limprecht R, Raschle NM, Vriends N, Trestman RL, Kirchner M, Kersten L. START NOW: a cognitive behavioral skills training for adolescent girls with conduct or oppositional defiant disorder - a randomized clinical trial. J Child Psychol Psychiatry. 2024 Mar;65(3):316-327. doi: 10.1111/jcpp.13896. Epub 2023 Oct 10. PMID 37814906